CLINICAL TRIAL: NCT00447681
Title: Ascending Single Dose Study of the Safety, Tolerability, Pharmacokinetiks, and Pharmacodynamics of ILV-094 Administered Intravenously and One Dose of ILV-094 Administered Subcutaneously to Healthy Subjects
Brief Title: Study of the Safety, Tolerability, Pharmacokinetics and Pharmcodynamics of ILV-094 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 3199K1-100
Record Dates: First submitted 2007-03-13; First posted 2007-03-15 (Estimated); Last update posted 2007-12-13 (Estimated); Status verified 2007-12

CONDITIONS: Healthy
MeSH Terms: interventions — fezakinumab

INTERVENTIONS:
Drug: ILV-094

SUMMARY:
This a randomized, double-blind placebo-controlled inpatient/outpatient, sequential group study of ascending single IV doses of ILV-094, an investigational drug, administered to healthy subjects. In addition, there will be one sub-cutaneous dose cohort, which will follow the 25 mg IV dose.

ELIGIBILITY:
* Healthy subjects (Men or women of nonchildbearing potential ), aged 18 to 50 years.
* Body mass index in the range of 18 to 30 Kg/m2 and body weight greater than 50 Kg.
* Healthy as determined by the investigator on the basis of medical history, physical examination, clinical laboratory test results, vital signs, and 12-lead electrocardiogram.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Estimated)
Dates: Start 2006-12; Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety, tolerability, pharmacokinetics and pharmcodynamics

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (1):
- Philadelphia, Pennsylvania, United States